CLINICAL TRIAL: NCT06869954
Title: Towards a More Standardized Bicuspid Aortic Valve Repair: Rationale and Design of CONTOUR Trial
Brief Title: Towards a More Standardized Bicuspid Aortic Valve Repair: Rationale and Design of CONTOUR Trial - a Randomized Trial
Acronym: CONTOUR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Augsburg (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); University Clinic Frankfurt (Other); Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-0625
Record Dates: First submitted 2025-01-22; First posted 2025-03-11 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Bicuspid Aortic Valve (BAV); Aortic Regurgitation Disease
Keywords: aortic regurgitation; aortic valve repair; annuloplasty; bicuspid aortic valve
MeSH Terms: conditions — Bicuspid Aortic Valve Disease; Aortic Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: CONTOUR is a prospective, randomized, parallel, two-arm, and assessor-blinded multicenter trial.
Who Masked: Outcomes Assessor
Masking Description: Because of the multicentre design, a MRI Core Center has been established to ensure standardized and rater-blinded analysis of the collected 4D flow MRI endpoints. To avoid any potential human bias, study-related radiologists (P.B., A.L.) at the MRI Core Center who are not involved in the treatment of study patients and are blinded to the group assignment will assess MRI-data in the specific MRI database separated from the main project eCRF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERNAL Group (Active Comparator): For the INTERNAL group, the HAART 200 internal annuloplasty ring (CorCym, London, UK), specifically designed for BAV morphology, will be used for all patients. Intraoperative sizing for the internal ring is based on the geometric orientation and size of the non-fused cusp. A standard ball sizer is used for the measurement of the non-fused cusp to assess commissural orientation and surface area of the non-fused cusp. Sizing typically results in values of 23mm or 25mm, with other sizes being very rare. Both commissural posts of the internal annuloplasty ring are fixed using two subcommissural sutures [10]. A modified technique for placement of transannular looping sutures will be used to secure the internal ring in the subannular position, as recently published [21]. Cusp maneuvers (i.e., shaving, thinning of the raphe, central plication sutures) will be performed to achieve an effective height of 8-10 mm. When indicated (i.e., for ascending aortic diameter > 45mm or aiming to achieve t
  Interventions: Device: Internal HAART 200 annuloplasty device
- EXTERNAL group (Active Comparator): For the EXTERNAL group, all study patients will undergo double external Dacron ring annuloplasty by simultaneous stabilization of the basal virtual ring and the STJ [22]. The surgical technique of double external annuloplasty, detailed by the Lansac group [22], involves aortic annulus sizing with a Hegar dilator to select the sizes of the external subannular annuloplasty ring and STJ ring (same size). After deep dissection of the aortic root, 6-7 2-0 pledgeted U sutures are placed circumferentially at the level of the virtual basal ring for external subannular ring implantation. Cusp maneuvers are performed similar to those in the INTERNAL group. STJ stabilization is achieved using an external STJ ring or ascending aortic replacement with a vascular tube graft (e.g., in cases with a high offspring of the right coronary artery). Treatment of the tubular ascending aorta is identical to the INTERNAL group.
  Interventions: Device: double external ring annuloplasty

INTERVENTIONS:
Device: Internal HAART 200 annuloplasty device — For the INTERNAL group, the HAART 200 internal annuloplasty ring (CorCym, London, UK), specifically designed for BAV morphology, will be used for all patients. Intraoperative sizing for the internal ring is based on the geometric orientation and size of the non-fused cusp. A standard ball sizer is used for the measurement of the non-fused cusp to assess commissural orientation and surface area of the non-fused cusp. Sizing typically results in values of 23mm or 25mm, with other sizes being very rare. Both commissural posts of the internal annuloplasty ring are fixed using two subcommissural sutures [10]. A modified technique for placement of transannular looping sutures will be used to secure the internal ring in the subannular position, as recently published [21]. Cusp maneuvers (i.e., shaving, thinning of the raphe, central plication sutures) will be performed to achieve an effective height of 8-10 mm. When indicated (i.e., for ascending aortic diameter > 45mm or aiming to achieve th
  Arms: INTERNAL Group
Device: double external ring annuloplasty — For the EXTERNAL group, all study patients will undergo double external Dacron ring annuloplasty by simultaneous stabilization of the basal virtual ring and the STJ [22]. The surgical technique of double external annuloplasty, detailed by the Lansac group [22], involves aortic annulus sizing with a Hegar dilator to select the sizes of the external subannular annuloplasty ring and STJ ring (same size). After deep dissection of the aortic root, 6-7 2-0 pledgeted U sutures are placed circumferentially at the level of the virtual basal ring for external subannular ring implantation. Cusp maneuvers are performed similar to those in the INTERNAL group. STJ stabilization is achieved using an external STJ ring or ascending aortic replacement with a vascular tube graft (e.g., in cases with a high offspring of the right coronary artery). Treatment of the tubular ascending aorta is identical to the INTERNAL group.
  Arms: EXTERNAL group

SUMMARY:
Background: Between one-third and one-half of patients with bicuspid aortic valve (BAV) disease develop significant aortic regurgitation (AR) at a young age, leading to cardiomyopathy and heart failure. Aortic valve repair is an evolving and still underused strategy in BAV patients with AR. The lack of sufficient standardization remains the main limitation of current repair techniques, resulting in an increased risk of AR recurrence and reoperation. The most controversial issue is the stabilization of the BAV annulus. The CONTOUR trial aims to compare two different BAV annuloplasty concepts in a prospective randomized study.

Methods: CONTOUR is a multicenter, randomized controlled trial designed to enroll 100 consecutive BAV patients with AR across four sites in Germany. BAV AR patients with an asymmetric configuration and without concomitant root aneurysm will be randomized 1:1 to undergo aortic valve repair using an internal HAART 200 annuloplasty device (i.e., INTERNAL group) (n=50) or external annuloplasty (i.e., double external ring annuloplasty) in the EXTERNAL group (n=50). 4D flow MRI will be performed preoperatively (t1), postoperatively at discharge (t2), and at 1-year follow-up (t3) for rater-blinded assessment of hemodynamic profiles (i.e., flow eccentricity) and regurgitation fraction at the MRI core-lab. Two hierarchically ordered primary endpoints will be considered: (1) postoperative reduction of flow eccentricity at hospital discharge and (2) regurgitation fraction (%) at 1-year follow-up.

Discussion: The CONTOUR trial is designed to test the hypothesis that an internal annuloplasty device, creating a completely symmetric post-repair BAV geometry, achieves superior aortic valve repair outcomes compared to external annuloplasty. If our hypothesis is confirmed, our study will significantly influence aortic valve repair practice and contribute to the refinement of guideline recommendations in the management of BAV patients with AR.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of fused BAV phenotype with an asymmetric configuration (commissural orientation < 170 degree) [14]
2. Severe aortic regurgitation (vena contracta (vc) > 6mm and/or pressure half-time (PHT) < 200 ms and/or effective regurgitant orifice area (EROA) > 30 mm2 and/or regurgitant volume (RV) > 60 ml/beat and/or left ventricular end-systolic diameter (LVESD) > 50mm (or indexed LVESD > 20mm/m2 BSA) and/or regurgitation fraction (RF) in cardiothoracic MRI > 40%) (at least one parameter is required) [15]
3. Isolated aortic valve surgery or concomitant procedure (including CABG and/or mitral/tricuspid valve surgery and/or ascending aortic surgery)
4. Willingness to participate and written informed consent
5. Age at surgery > 18 years

Exclusion Criteria:

1. Moderate/severe BAV stenosis (pmean > 20mmHg)
2. Moderate/severe BAV cusp calcifications extending beyond the raphe region and/or necessitating patch implantation (deemed irreparable based on preoperative TOE (as by decision of the operating surgeon)
3. Concomitant aortic root aneurysm > 45mm requiring simultaneous aortic root surgery [16]
4. Acute/subacute BAV endocarditis
5. Contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Post-repair reduction of flow eccentricity in percent assessed via cardiac magnetic resonance imaging (MRI) | Between the preoperative baseline (max. 30 days preoperative) (t1) and postoperative (pre-discharge) (t2) periods
  Flow eccentricity (in percent) will be assessed using cardiac with phase-contrast imaging. Flow eccentricity is calculated based on the deviation of the flow jet from the center of the vessel lumen. Measurements will be performed pre- and post-repair to determine the percentage reduction in flow eccentricity. Measurements will be performed pre- and post-repair to determine the percentage reduction in flow eccentricity.
Regurgitation fraction in percent assessed via cardiac magnetic resonance imaging (CMR) | Measurements will be taken at baseline (t1), an early post-operative time point (t2), and at 1-year follow-up (t3). The primary analysis will assess changes from baseline (t1) to both post-operative time points (t2 and t3).
  The regurgitation fraction (%) will be assessed using cardiac magnetic resonance imaging (CMR) with phase-contrast imaging. Regurgitation fraction is calculated as the percentage of retrograde blood flow relative to the total blood flow through the valve. Measurements will be performed at baseline (pre-repair) and after the intervention (post-repair) to evaluate changes in regurgitation fraction.
  For the second primary endpoint (regurgitation fraction), the dependent variable is the post (t2 and t3) value. The study group, time post-surgery (t2 and t3), the interaction between the study group and time post-surgery measurement, and center are included as independent fixed-effect variables.

SECONDARY OUTCOMES:
Severity of aortic regurgitation (mild/moderate/severe)* | Assessment at month 6 (t2) and month 12 (t3) in both study groups
  Severity will be assessed at months 6 (t2) and 12 (t3) in both study groups. The assessment is based on clinical imaging data, including transthoracic echocardiography (TTE) and cardiac MRI as available.
Transvalvular gradient (mmHg) | Assessment at month 6 (t2) and month 12 (t3) in both study groups
All-cause mortality (yes/no) | Assessment at month 6 (t2) and month 12 (t3) in both study groups
Adverse cardiac events (MACCE) (yes/no) | Assessment at month 6 (t2) and month 12 (t3) in both study groups
Aortic valve re-intervention (yes/no) | Assessment at month 6 (t2) and month 12 (t3) in both study groups
Re-hospitalization due to cardiac reasons (yes/no) | Assessment at month 6 (t2) and month 12 (t3) in both study groups
Device-related complications (safety endpoint) (yes/no) | Assessment at month 6 (t2) and month 12 (t3) in both study groups
Assessment of valvular cardiomyopathy: LV diameters (LVESD, LVEDD) | Assessment at post-procedural baseline (Day 0 = t1), month 6 (t2), and month 12 (t3) in both study groups.
  Left ventricular end-systolic diameter (LVESD) and left ventricular end-diastolic diameter (LVEDD) measured by echocardiography and/or cardiac MRI.
Assessment of valvular cardiomyopathy LV volumes (LVESV, LVEDV) | Assessment at post-procedural baseline (t1), month 6 (t2), and month 12 (t3) in both study groups.
  Left ventricular end-systolic volume (LVESV) and left ventricular end-diastolic volume (LVEDV) measured by echocardiography and/or cardiac MRI.
Assessment of valvular cardiomyopathy LV strain (GLS) | Assessment at post-procedural baseline (t1), month 6 (t2), and month 12 (t3) in both study groups.
  Global longitudinal strain (GLS) of the left ventricle assessed by echocardiography and/or cardiac MRI.

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - University Hospital Augsburg, Augsburg, Bavaria
  - University Heart and Vascular Center Frankfurt, Frankfurt am Main, Hesse
  - Heart Center Leipzig, Leipzig, Saxony
  - Medical Center Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Girdauskas E, Stock S, Hofbauer D, Petersen J, Reichenspurner H, Holubec T, Walther T, Vogl T, Borger M, Gutberlet M, Kroncke T, Decker J, Zapf A, Lezius S, Lenz A, Lansac E, Bannas P. Towards a More Standardized Bicuspid Aortic Valve Repair: Rationale and Design of the CONTOUR Trial. Eur J Cardiothorac Surg. 2025 Dec 1;67(12):ezaf360. doi: 10.1093/ejcts/ezaf360. PMID 41124604